CLINICAL TRIAL: NCT00491621
Title: Study Evaluating the Interest of Cytology-molecular Tumor Markers Association for the Diagnostic Strategy in Adult Kidney Tumors
Brief Title: Evaluation of Diagnostic Value of Molecular Markers in Renal Cancer
Acronym: CMM
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: No enough inclusion. The aim is no longer relevant. The sponsor decided to stop this study.
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 0501106
Record Dates: First submitted 2007-06-25; First posted 2007-06-26 (Estimated); Last update posted 2015-06-04 (Estimated); Status verified 2015-06

CONDITIONS: Kidney Neoplasms
Keywords: kidney; tumor; Molecular Markers; Cytology; Histology; Cystic kidney tumor
MeSH Terms: conditions — Kidney Neoplasms; Neoplasms | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Other): surgery or biopsy of the kidney tumor
  Interventions: Procedure: surgery or biopsy of the kidney tumor

INTERVENTIONS:
Procedure: surgery or biopsy of the kidney tumor — surgery or biopsy of the kidney tumor

SUMMARY:
Renal cancer is frequent and its diagnosis mainly dependant on imaging. More than 50% of renal tumors are currently diagnosed without symptoms. However, 20% of small solid tumors are benign and this percentage is much higher in atypical cystic tumors Bosniak II and III, where 76% and 59% are benign respectively. Determining the malignancy by imaging in these cases is difficult and sometimes impossible. The fine needle aspiration (FNA) cytology or biopsy is necessary. The diagnostic sensitivity and specificity with biopsy are high, but the potential tumor contamination is a major risk. The FNA cytology is simple and safe, but its sensitivity is about 50%. We are conducting a multicentric prospective study to add the molecular markers in FNA cytology as a new diagnostic method in imaging-indeterminate renal tumors.

Four molecular markers including MN/CA9, vimentin, KIT, and S100A1 will be studied. These four markers have been reported to have a differential diagnostic value in renal tumors. MN/CA9 and vimentin are often found in conventional renal cancers. KIT is frequently expressed in renal oncocytomas and chromophobe renal cancers. S100A1 may further distinguish renal oncocytoma from chromophobe renal cancer. These markers will be analyzed by real time polymerase chain reaction (RT-PCR).

The aim of this study is to evaluate the diagnostic performance of the association cytology-molecular markers in imaging-indeterminate renal tumors (small solid tumors and cystic tumors ≥ Bosniak III). About 156 patients will be included in five French clinical centers including Saint-Etienne, Marseille, Grenoble, Toulouse, and Nancy.

The expected results will improve the preoperative diagnostic accuracy in renal tumors.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of kidney tumor < 4 cm
* Cystic kidney tumor (Bosniak > IIF)
* Consent signed

Exclusion Criteria:

* Benign tumor confirmed
* Impossibility to do abdominal pelvic ultra-sound or abdominal thoracic scanner
* Contraindication for renal puncture

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2007-04; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Histologic diagnostic (tumor) | after surgery or biopsy

SECONDARY OUTCOMES:
Cytology-molecular tumor markers association diagnostic (tumor) | after surgery or biopsy
Molecular tumor markers association diagnostic (blood + urine) | 3, 6, 9, 12, 15, 18, 21 and 24 months after biopsy

CONTACTS AND LOCATIONS:
Overall Officials: Jacques TOSTAIN, PhD-MD, Study Chair — CHU de Saint-Etienne
Locations (7):
- France (7):
  - CHU de Grenoble, Grenoble
  - Hospices Civils de Lyon - Edouard Herriot, Lyon
  - AP-HM Hôpital Nord, Marseille
  - AP-HM Hôpital Salvator, Marseille
  - CHU de Nancy, Nancy
  - CHU de Saint-Etienne, Saint-Etienne
  - CHU de Toulouse, Toulouse

REFERENCES:
- [Background] Li G, Cuilleron M, Cottier M, Gentil-Perret A, Lambert C, Genin C, Tostain J. The use of MN/CA9 gene expression in identifying malignant solid renal tumors. Eur Urol. 2006 Feb;49(2):401-5. doi: 10.1016/j.eururo.2005.10.025. Epub 2005 Dec 19. PMID 16387417
- [Background] Li G, Cuilleron M, Gentil-Perret A, Cottier M, Passebosc-Faure K, Lambert C, Genin C, Tostain J. Rapid and sensitive detection of messenger RNA expression for molecular differential diagnosis of renal cell carcinoma. Clin Cancer Res. 2003 Dec 15;9(17):6441-6. PMID 14695146
- [Background] Li G, Barthelemy A, Feng G, Gentil-Perret A, Peoc'h M, Genin C, Tostain J. S100A1: a powerful marker to differentiate chromophobe renal cell carcinoma from renal oncocytoma. Histopathology. 2007 Apr;50(5):642-7. doi: 10.1111/j.1365-2559.2007.02655.x. PMID 17394501
- [Background] Li G, Feng G, Gentil-Perret A, Genin C, Tostain J. CA9 gene expression in conventional renal cell carcinoma: a potential marker for prediction of early metastasis after nephrectomy. Clin Exp Metastasis. 2007;24(3):149-55. doi: 10.1007/s10585-007-9064-z. Epub 2007 Mar 28. PMID 17390110
- [Background] Li G, Gentil-Perret A, Lambert C, Genin C, Tostain J. S100A1 and KIT gene expressions in common subtypes of renal tumours. Eur J Surg Oncol. 2005 Apr;31(3):299-303. doi: 10.1016/j.ejso.2004.11.009. PMID 15780567